CLINICAL TRIAL: NCT01374737
Title: ED50 of Dexmedetomidine for Reduction of Emergence Agitation Incidence Undergoing Tonsillectomy or Adenoidectomy in Desflurane Anesthesia Following Sevoflurane Induction in Children
Brief Title: ED50 of Dexmedetomidine to Prevent Emergence Agitation in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Hee-Soo Kim, SNUH
Allocation: Non-Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KHS_1
Record Dates: First submitted 2011-06-09; First posted 2011-06-16 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Agitation
MeSH Terms: conditions — Psychomotor Agitation | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- dexmedetomidine, children (Other)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — dexmedetomidine, 0.1ug/kg up or down
  Other Names: precedex

SUMMARY:
There are several recommended doses of dexmedetomidine for prevention of emergence agitation in children. In this study, the investigators examine ED50 in prevention of emergence agitation after tonsillectomy or adenoidectomy in children.

DETAILED DESCRIPTION:
To investigate ED50, Dixon's up and down method will be used.

ELIGIBILITY:
Inclusion Criteria:

* tonsillectomy or adenoidectomy

Exclusion Criteria:

* recent URI

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2011-06; Primary Completion 2011-12 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
agitation | 30 minutes

SECONDARY OUTCOMES:
pain | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Soo Kim, M.D, PhD, Study Director — Seoul National University Hospital
Locations (1):
- SNUH, Seoul, South Korea